CLINICAL TRIAL: NCT04143997
Title: Diastolic Dysfunction PPCM in Patients With Documented Left Ventricular Systolic Function Recovery
Status: Withdrawn | Type: Observational
Why Stopped: No pt enrolled
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Other Study IDs: PRO00036227
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Peripartum Cardiomyopathy; Diastolic Dysfunction
MeSH Terms: conditions — Peripartum Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PPCM with Diastolic Dysfunction & Normal Systolic Function: The patient population examined will include patients diagnosed with peripartum cardiomyopathy who have diastolic dysfunction and normal systolic function.
  Interventions: Diagnostic Test: A clinical Transthoracic echocardiogram

INTERVENTIONS:
Diagnostic Test: A clinical Transthoracic echocardiogram — A previously clinically completed transthoracic echocardiogram will be utilized to assess for diastolic dysfunction in the presence of normal systolic function for patients with previously diagnosed peripartum cardiomyopathy.

SUMMARY:
The purpose of this project is to evaluate parameters of diastolic dysfunction assessed by clinical echocardiogram in patients who have had recovery of systolic function.

ELIGIBILITY:
Inclusion Criteria:

1. Female.
2. Greater than age 18 years at the time of peripartum cardiomyopathy diagnosis.
3. Adults with a current or prior diagnosis of peripartum cardiomyopathy and documented recovered of left ventricular systolic function.
4. Documented recovered of LV systolic performance defined as LVEF > 50%.

Exclusion Criteria:

1. No pregnancy history.
2. No diagnosis of peripartum cardiomyopathy.
3. Non-recovery of LV systolic function.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a current or prior diagnosis of peripartum cardiomyopathy and documented recovered of left ventricular systolic function.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-01-29 (Estimated); Study Completion 2021-01-29 (Estimated)

PRIMARY OUTCOMES:
Report the incidence of diastolic dysfunction in peripartum cardiomyopathy patients with full systolic function recovery | January 1, 2014 through September 1, 2019
  Investigators will review and report incidence of remaining diastolic dysfunction for local patient population which have recovered systolic function.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Thordsen, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States